CLINICAL TRIAL: NCT05168982
Title: Development of Fully Automated Non-Invasive MRI Applications for Diagnosis and Staging of Liver Fibrosis and Inflammation
Brief Title: Development of Non-Invasive MRI Applications for Liver Fibrosis and Inflammation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chen Weitian, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2021.372
Record Dates: First submitted 2021-12-10; First posted 2021-12-23 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Liver Fibrosis
Keywords: MRI, liver fibrosis, liver inflammation
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Chronic liver disease (CLD) patients at stage A0 of liver inflammation
- Chronic liver disease (CLD) patients at stage A1 of liver inflammation
- Chronic liver disease (CLD) patients at stage A2 of liver inflammation
- Chronic liver disease (CLD) patients at stage A3 of liver inflammation
- Chronic liver disease (CLD) patients at stage F0 of liver fibrosis
- Chronic liver disease (CLD) patients at stage F1 of liver fibrosis
- Chronic liver disease (CLD) patients at stage F2 of liver fibrosis
- Chronic liver disease (CLD) patients at stage F3 of liver fibrosis
- Chronic liver disease (CLD) patients at stage F4 of liver fibrosis
- healthy subjects

SUMMARY:
Chronic liver disease is a major healthcare problem in Hong Kong and worldwide. The diagnosis of liver fibrosis and inflammation in patients with chronic liver disease has important prognostic and therapeutic implications. The current gold standard to evaluate and stage the severity of liver fibrosis and inflammation is based on liver biopsies, which are invasive and impractical for screening and monitoring the disease. The existing non-invasive methods still have significant limitations to meet the challenge.

Magnetic resonance effect can be used to obtain the molecular-level information on the biochemical properties of human tissues. The investigators will develop non-invasive quantitative MRI technologies to evaluate and stage liver fibrosis and inflammation. Our approaches are based on the endogenous contrast mechanism and thus do not need to inject an MRI contrast agent. Our approaches can be implemented on a regular MRI scanner and do not need any extra hardware. To enable the technology for routine clinical use, the investigators will develop fully automated post-processing techniques for the proposed MRI acquisition approaches. The investigators will perform multi-center clinical studies in Hong Kong and mainland China to validate our imaging measurements by histopathologic results from liver biopsies on patient cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 18 and 65.
* Chronic liver disease (CLD) patients at different stages of liver inflammation (A0-3) and liver fibrosis (F0-4).
* CLD patients who have indications and are scheduled to undergo liver biopsy.

Exclusion Criteria:

* Patients diagnosed with HCC or other types of cancers.
* Patients who had undergone liver transplantation before enrollment.
* Any contraindications to either liver biopsy or MRI scan.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic liver disease (CLD) patients at different stages of liver inflammation (A0-3) and liver fibrosis (F0-4)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare the measurement between subjects with different grades of liver inflammation and stages of liver fibrosis | one year
  T-Test or one-way analysis of variance (ANOVA) will be performed for continuous variables with normally distribution, along with Kruskal-Wallis test or Mann-Whitney U test for continuous variables with skewed or unknown distribution, while χ2 or Fisher exact test will be carried out for categorical variables.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Prince of Wale Hospital, Hong Kong, Shatin, Hong Kong